CLINICAL TRIAL: NCT01882712
Title: Phase 3 Efficacy and Safety Study of CD07805/47 Topical Gel in Subjects With Persistent Facial Erythema
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.03.SPR.40191
Record Dates: First submitted 2013-06-14; First posted 2013-06-20 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Erythema
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CD07805/47 Gel 0.5% (Experimental): active arm
  Interventions: Drug: CD07805/47 Gel 0.5%
- CD07805/47 Gel Placebo (Placebo Comparator): Comparator arm
  Interventions: Drug: CD07805/47 Gel Placebo

INTERVENTIONS:
Drug: CD07805/47 Gel 0.5%
  Arms: CD07805/47 Gel 0.5%
Drug: CD07805/47 Gel Placebo
  Arms: CD07805/47 Gel Placebo

SUMMARY:
The purpose of this study is to compare the efficacy and assess the safety of CD07805/47 gel 0.5% applied topically once daily for 29 days versus vehicle control, in subjects with moderate to severe chronic persistent vascular facial erythema

ELIGIBILITY:
Inclusion Criteria:

* Male or female, who is at least 18 years of age or older at screening visit.
* Presence of chronic persistent vascular facial erythema for ≥ 3 months by history.
* A Clinician's Erythema Assessment (CEA) score of ≥3 at Screening and at Pre-dose (T0) on Baseline/Day 1.
* A Patient Self Assessment (PSA) score of ≥3 at Screening and at Pre-dose (T0) on Baseline/Day 1.

Exclusion Criteria:

* More than 2 facial inflammatory lesions (papules, pustules, and nodules).
* Presence of areas of significant scaling or crusting on the face.
* Presence of psoriatic lesions on the face.
* Presence of any other dermatological condition of the face that, in the opinion of the Investigator, may significantly interfere with the interpretation of the clinical trial results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Composite success on both CEA (Clinician Erythema Assessment ) and PSA (Patient Self Assessment) | Day 29
  2-grade improvement on both CEA and PSA at Hours 3, and 6 after Pre-dose (T0)on Day 29

SECONDARY OUTCOMES:
Composite improvement on both CEA (Clinician Erythema Assessment ) and PSA (Patient Self Assessment) | Day 1
  1-grade improvement on both CEA and PSA at 30 minutes after pre-dose (T0) on Day 1